CLINICAL TRIAL: NCT04998643
Title: Muscle Catabolism and Its Impact on Functional Outcomes in Children Following Cardiac Surgery
Brief Title: Muscle Catabolism and Outcomes in Children Following Cardiac Surgery
Acronym: MOCHI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: Academy of Nutrition and Dietetics (Other)
Responsible Party: Principal Investigator, Kimberly I. Mills, MD, Staff Physician, Boston Children's Hospital
Other Study IDs: IRB-P00038896
Record Dates: First submitted 2021-07-19; First posted 2021-08-10 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Congenital Heart Disease; ICU Acquired Weakness; Catabolic State
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Muscle ultrasound to estimate lean body mass — The investigators will perform serial muscle ultrasounds in the postoperative period to estimate lean body mass.

SUMMARY:
Background & Significance. Children with congenital heart disease (CHD) have experienced improved postoperative survival shifting the focus away from minimizing mortality to curtailing morbidities. Critical illness following cardiac surgery induces catabolism which may impact functional status. Catabolism, a state in which protein breakdown exceeds protein synthesis, can lead to lean body mass (LBM) breakdown. LBM loss has been associated with poor clinical outcomes. Muscle ultrasound (mUS) has been utilized to measure LBM changes and the functional status score (FSS) was developed to assess functional status changes in children following hospitalization. The ability to identify LBM loss acutely and its association with FSS changes may lead to earlier interventions to preserve LBM and aid in outcome prediction.

Specific Aims & Hypotheses. Specific Aim 1 is to identify the percent change in LBM by mUS during the first postoperative week in children following complex cardiac surgery. Specific Aim 2 is to evaluate the relationship between percent change in LBM during the first postoperative week and the FSS at discharge and 6 and 12-month follow-up in children with CHD following complex cardiac surgery. The investigators hypothesize children with CHD following complex cardiac surgery will experience a decline in LBM and that there is a direct relationship between the change in LBM and postoperative FSS follow-up.

Study Design & Methods. The investigators are conducting a single-center, prospective, observational cohort study. Consecutive children (> 3 months and < 18 years of age) with CHD undergoing biventricular conversion will be enrolled. Patients will undergo a baseline mUS and FSS at the time of the index operation. Interval mUS will be obtained on the third and seventh postoperative day. Discharge mUS and FSS will be obtained and a remote FSS will be requested by the family at 6 and 12-months postoperatively. Demographics, pertinent laboratory, concomitant medications, nutrition and ultrasound variables will be collected.

Outcomes. The primary outcomes will be change in LBM during the first postoperative week and change in FSS at 6 and 12-month follow-up in children following complex cardiac surgery. Change in LBM will be defined as a percent change in cross-sectional area of the quadriceps muscle layer thickness (QMLT). Change in FSS will be significant if the score drops 3 points or more from baseline at postoperative follow-up.

DETAILED DESCRIPTION:
The central objective of our single center, pilot study in children with CHD following cardiac surgery is to identify serial changes in QMLT, as an estimate of LBM, during the first postoperative week, and to examine its relationship to functional status, assessed by FSS, after hospital discharge.

Primary Aim 1. To measure the percent change in QMLT by mUS during the first postoperative week in children undergoing complex cardiac surgery. The investigators hypothesize children undergoing complex cardiac surgery will have a mean decline of at least 10% in QMLT during the first postoperative week.

Primary Aim 2. To examine the relationship between percent change in QMLT during the first postoperative week and FSS at 3 and 6-months. The investigators hypothesize there is a direct relationship between percent change in QMLT during the first postoperative week and FSS at 3 and 6-months following surgery.

Secondary Aim 1. To explore the relationship between nitrogen balance, defined as the difference between total nitrogen intake and total urinary nitrogen loss, and mean change in QMLT during the first postoperative week. The investigators hypothesize there is a direct correlation between nitrogen balance and mean change in QMLT during the first postoperative week in children following complex cardiac surgery.

The proposed utilization of mUS to measure alterations in body composition during the acute phase of critical illness may provide early prediction of subsequent functional status decline.

ELIGIBILITY:
Inclusion Criteria:

1. children > 3 months and < 18 years old,
2. diagnosed with CHD, and
3. undergoing biventricular conversion.

Exclusion Criteria:

1. diagnosis of muscular dystrophy or myopathy,
2. lower extremity injury or infection during the current hospitalization,
3. enrolled in a concurrent nutritional intervention trial, or
4. admitted for palliative care.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with congenital heart disease admitted to the cardiac intensive care unit following complex cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in lean body mass | 7 days postoperatively
  The investigators are measuring the change in lean body mass estimated by quadriceps muscle layer thickness (QMLT)
Change in functional status | 6 and 12 months
  The investigators will measure functional status at 6 and 12-month follow-up to investigate the association between change in QMLT and functional status

SECONDARY OUTCOMES:
Relationship of nitrogen balance to lean body mass changes | 12-24 hours postoperatively
  The investigators will measure urinary nitrogen balance to investigate its relationship to mean change in QMLT during the first postoperative week

CONTACTS AND LOCATIONS:
Overall Officials: Lori Bechard, RD, PhD, Study Director — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared with other researchers.